CLINICAL TRIAL: NCT04544618
Title: Preoperative Virtual Reality for Cancer Surgery Patients: A Feasibility and Pilot Study
Brief Title: Evaluation of a Pre-surgical Virtual Reality Simulation for Cancer Surgery Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Jordana Sommer, Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: HS23957 (H2020:247); 322523 340300 2000 (Other Grant/Funding Number: New Frontiers)
Record Dates: First submitted 2020-08-19; First posted 2020-09-10 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Anxiety State
Keywords: Preoperative anxiety; Cancer; Virtual reality; Feasibility; Pilot study
MeSH Terms: conditions — Anxiety Disorders; Neoplasms

STUDY DESIGN:
Intervention Model Description: This study will employ a single-blind randomized design (1:1 randomization; stratified according to surgery type [with vs. without reconstruction] and whether or not neoadjuvant chemotherapy was received; stratification will designate equal proportions of participants with these characteristics across each of the two study groups).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will be exposed to a virtual reality simulation of the operating room environment for a minimum of ten minutes.
  Interventions: Device: Virtual reality operating room simulation
- Treatment as usual group (No Intervention): Participants will receive standard of care with no additional intervention aside from information received at their surgical oncology appointment and optional preoperative education classes (available to all patients).

INTERVENTIONS:
Device: Virtual reality operating room simulation — The virtual reality simulation will begin with the participant sitting on a hospital bed wearing the virtual reality headset and holding the controllers. Participants will be oriented to the environment and provided with an explanation of how to navigate through the simulation (for approximately 2 minutes). Next, participants will explore the virtual operating room for a minimum of 5 minutes, or longer if desired. Following the exploration period, the scripted portion of the simulation will be begin. Here, participants will be taken through the mock anesthetic induction process (the virtual anesthetist will speak to the patient and walk them through the steps and the virtual nurse will assist). The simulation ends after the virtual oxygen mask is placed over the participant's mouth and the screen darkens.
  Arms: Intervention group

SUMMARY:
This study will pilot test and explore the feasibility of a virtual reality simulation of the operating room environment to reduce anxiety/distress in cancer surgery patients. Study objectives are to evaluate recruitment and data collection procedures, outcome measures, participant feedback on the virtual reality operating room intervention, and the inclusion of a treatment as usual group, and effects of the intervention on symptoms of anxiety/distress. Results of this study will inform the design of an upcoming larger-scale RCT to assess the efficacy of this intervention

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18
* Can speak and read English
* Has a cancer diagnosis
* Scheduled/being scheduled to undergo cancer surgery under general anesthesia at the Health Sciences Centre (Winnipeg, MB)

Exclusion Criteria:

* Those who do not meet any inclusion criteria
* Those who are not competent to provide informed consent (e.g., due to cognitive impairment)
* Those who are unable to participate in a virtual reality intervention (e.g., due to visual/auditory impairment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Self-reported impressions of the virtual reality operating room simulation | Baseline
  Patient acceptability questionnaire with open and close-ended items assessing patients' impressions of the intervention
Self-reported impressions of the virtual reality operating room simulation | 5 days
  Patient acceptability questionnaire with open and close-ended items assessing patients' impressions of the intervention

SECONDARY OUTCOMES:
NCCN Distress Thermometer | Baseline, up to 2 weeks after baseline on day of scheduled surgery, 5 days, and 30 days
  VAS self-reported distress on a scale of 0-10
NCCN Anxiety Thermometer | Baseline, up to 2 weeks after baseline on day of scheduled surgery, 5 days, and 30 days
  VAS self-reported anxiety on a scale of 0-10
iGroup Presence Questionnaire | Immediately after the intervention
  Assessing the sense of presence experienced by participants in the virtual environment
Preoperative Intrusive Thoughts Inventory (PITI) | Baseline and up to 2 weeks after baseline on day of scheduled surgery
  PITI questionnaire
Amsterdam Preoperative Anxiety Information Scale (APAIS) | Baseline and up to 2 weeks after baseline on day of scheduled surgery
  APAIS questionnaire

OTHER OUTCOMES:
PROMIS emotional distress- anxiety | Baseline, 5 days, and 30 days
  PROMIS anxiety questionnaire
PROMIS emotional distress- depression | Baseline, 5 days, and 30 days
  PROMIS depression questionnaire
PROMIS global health | Baseline, 5 days, and 30 days
  PROMIS global health questionnaire
PROMIS fatigue | Baseline, 5 days, and 30 days
  PROMIS fatigue questionnaire
PROMIS emotional support | Baseline, 5 days, and 30 days
  PROMIS emotional support questionnaire
PROMIS pain intensity | 5 days and 30 days
  PROMIS pain intensity questionnaire
Peritraumatic Distress Inventory (PDI) | Baseline and 5 days
  PDI questionnaire
Primary Care PTSD Screen for DSM-5 (PC-PTSD-5) | Baseline and 30 days
  PC-PTSD-5 questionnaire
Brief Resilient Coping Scale (BRCS) | Baseline, 5 days, and 30 days
  BRCS questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jordana Sommer, MA, Principal Investigator — University of Manitoba; Renée El-Gabalawy, PhD, Principal Investigator — University of Manitoba; Kristin Reynolds, PhD, Study Director — University of Manitoba; Pamela Hebbard, MD, Study Director — University of Manitoba; Natalie Mota, PhD, Study Director — University of Manitoba; Alan Mutch, MD, Study Director — University of Manitoba; Thomas Mutter, MD, Study Director — University of Manitoba; Rakesh Arora, MD, Study Director — University of Manitoba; Jessica Maples-Keller, PhD, Study Director — Emory University
Locations (1):
- Health Sciences Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Gabalawy R, Sommer JL, Hebbard P, Reynolds K, Logan GS, Smith MSD, Mutter TC, Mutch WA, Mota N, Proulx C, Gagnon Shaigetz V, Maples-Keller JL, Arora RC, Perrin D, Benedictson J, Jacobsohn E. An Immersive Virtual Reality Intervention for Preoperative Anxiety and Distress Among Adults Undergoing Oncological Surgery: Protocol for a 3-Phase Development and Feasibility Trial. JMIR Res Protoc. 2024 May 14;13:e55692. doi: 10.2196/55692. PMID 38743939
- [Derived] Sommer JL, Reynolds K, Hebbard P, Smith MSD, Mota N, Mutch WAC, Maples-Keller J, Roos L, El-Gabalawy R. Preoperative Virtual Reality to Expose Patients With Breast Cancer to the Operating Room Environment: Feasibility and Pilot Case Series Study. JMIR Form Res. 2024 Jan 17;8:e46367. doi: 10.2196/46367. PMID 38231570